CLINICAL TRIAL: NCT01232348
Title: Symbicort Turbuhaler 30/60 Clinical Experience Investigation
Acronym: SURE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589IL00001
Record Dates: First submitted 2010-10-31; First posted 2010-11-02 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma; Symbicort
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symbicort: Those with an exposure

SUMMARY:
The purpose of this study is to confirm the safety (ADR related to beta stimulant drugs, unexpected ADRs) and efficacy of Symbicort in daily practice and the control status on bronchial asthma and Patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Symbicort for the first time due to bronchial asthma

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Symbicort for the first time due to bronchial asthma
Sampling Method: Non-Probability Sample
Enrollment: 3643 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Range of 12 weeks

SECONDARY OUTCOMES:
The level of asthma control | Range of 12 weeks
The level of patient satisfaction with Symbicort | Range of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshida Shigeru, MD, Study Director — AstraZeneca
Locations (47):
- Japan (47):
  - Research Site, Okazaki, Aichi-ken
  - Research Site, Akita, Akita
  - Research Site, Aomori, Aomori
  - Research Site, Chiba, Chiba
  - Research Site, Ehime, Ehime
  - Research Site, Fukui-shi, Fukui
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Fukushima, Fukushima
  - Research Site, Gifu, Gifu
  - Research Site, Gunma, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Hokkaido, Hokkaido
  - Research Site, Hyogo, Hyōgo
  - Research Site, Ibaraki, Ibaraki
  - Research Site, Ishikawa, Ishikawa-ken
  - Research Site, Numakunai, Iwate
  - Research Site, Kagawa, Kagawa-ken
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kanagawa, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Miemachi, Mie-ken
  - Research Site, Miyagi, Miyagi
  - Research Site, Miyazaki, Miyazaki
  - Research Site, Nagano, Nagano
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Nara, Nara
  - Research Site, Niigata, Niigata
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Okayama, Okayama-ken
  - Research Site, Okinawa, Okinawa
  - Research Site, Osaka, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Saitama, Saitama
  - Research Site, Shiga, Shiga
  - Research Site, Shimane, Shimane
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Tochigi, Tochigi
  - Research Site, Tokushima, Tokushima
  - Research Site, Tokyo, Tokyo
  - Research Site, Tottori-shi, Tottori
  - Research Site, Toyama, Toyama
  - Research Site, Wakayama, Wakayama
  - Research Site, Yamagata, Yamagata
  - Research Site, Yamaguchi, Yamaguchi
  - Research Site, Yamanashi, Yamanashi